CLINICAL TRIAL: NCT03377764
Title: Can Anesthesia Trainees Effectively Use Ultrasound Imaging to Facilitate the Performance of Spinal Anesthesia in Patients With Poorly-palpable Surface Landmarks?
Brief Title: Spinal Anesthesia in Patients With Poorly-palpable Surface Landmarks
Status: Terminated | Type: Observational
Why Stopped: The interim data analysis shows no significant difference between groups
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 11-0054-A
Record Dates: First submitted 2016-10-31; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2011-05

CONDITIONS: Regional Anesthesia
Keywords: Spinal Anesthetic,; Ultrasound guided Neuroaxial block,; Anesthesia Trainees

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Landmark Technique: Control group
  Interventions: Procedure: Landmark Technique Control group
- Ultrasound guided technique: Neuroaxial block using Ultrasound guidance
  Interventions: Procedure: Neuroaxial block using Ultrasound Guidance

INTERVENTIONS:
Procedure: Landmark Technique Control group — Spinal Anesthetic
  Groups: Landmark Technique
Procedure: Neuroaxial block using Ultrasound Guidance — Ultrasound guided Spinal Anesthetic
  Groups: Ultrasound guided technique

SUMMARY:
Anesthesia trainees can perform spinal anesthesia in patients who have poorly-palpable surface landmarks with fewer needle passes using an ultrasound-guided technique compared to the conventional surface landmark-guided technique.

DETAILED DESCRIPTION:
Neuraxial blockade has traditionally been accomplished using a surface landmark-guided technique, in which the approximate location of the neuraxial midline, lumbar interspinous and interlaminar spaces are determined based on palpation of the intercristal line and the tips of the spinous processes. It is not surprising, therefore, that the technical difficulty of neuraxial blockade (usually measured in terms of the number of needle passes required for success) correlates with the quality of palpable surface landmarks.

Reducing the technical difficulty of neuraxial blockade is desirable as multiple needle insertion attempts may increase the risk of complications such as post-dural puncture headache, paresthesiae, and epidural hematoma. Ultrasound (US) imaging of the spine can help in this regard by more precisely identifying landmarks, determining the intervertebral level, and measuring the depth to the epidural space. It has been shown to facilitate the performance of neuraxial block in the obstetric population, and our group has also demonstrated similar benefits in the older non-obstetric population. In a feasibility study of US-guided spinal anesthesia for total joint replacement surgery, achieved successful spinal anesthesia with a single needle insertion attempt in 84% of these patients, despite the fact that nearly half of them had poorly palpable surface landmarks.This compares well with large prospective cohort studies which report successful neuraxial blockade on the first needle insertion attempt in 61-64% of all patients. Investigators recently completed a randomized controlled trial in which 120 patients with difficult anatomical landmarks (defined as poorly palpable surface landmarks and a BMI>35 kgm-2, significant spinal deformity, or spinal surgery resulting in distortion or absence of surface landmarks) received spinal anesthesia performed by experienced anesthesiologists using either a conventional surface landmark-guided technique or an US-guided technique. There was a two-fold difference between the US-guided group and the control group in the first-attempt success rate (62% vs 32%, P<0.001), and the median number of needle passes required for success (6 vs 13, P=0.003).

The main limitation of all clinical studies conducted to date on US-guided neuraxial block is that ultrasound imaging was performed solely by experienced operators; although in two studies the neuraxial block itself (but not the ultrasound scan) was performed by trainees.

Investigators believe that the benefits of the US-guided technique can be realized when it is performed in its entirety by novices, e.g. anesthesia trainees. Investigators therefore designed this study to establish if novices are able to use the US-guided technique to facilitate the performance of spinal anesthesia in obese patients with poorly-palpable landmarks.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for elective total hip or knee replacement under spinal anesthesia who have poorly palpable or impalpable spinous processes
* BMI ≥ 35 kgm-2

Exclusion Criteria:

* Inability or refusal to provide informed consent,
* Bleeding diathesis,
* Allergy to local anesthetics
* Contra-indication to spinal anesthesia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will recruit patients presenting for elective total hip or knee replacement under spinal anesthesia, who have poorly palpable or impalpable spinous processes and a body mass index (BMI) ≥ 35 kgm-2. Exclusion criteria include inability or refusal to provide informed consent, bleeding diathesis, allergy to local anesthetics, or any other contra-indication to spinal anesthesia. Criteria for withdrawal after enrolment will include cancellation of surgery, unavailability of personnel with the requisite experience to perform the ultrasound-guided technique, and patient refusal to participate or continue with the study at any point up to completion of the US scan.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The rate of successful dural puncture on the first needle insertion attempt. | 2012-2013
  Insertion attempts are defined as complete withdrawal of the needle or introducer from the skin followed by re-insertion, and are distinguished from redirection attempts, which are defined as changes in needle trajectory that do not involve complete withdrawal of the needle from the skin. 1,2.14,15 This will be assessed by two blinded observers from an anonymized video recording of the operator's hands as they perform the spinal anesthetic.

SECONDARY OUTCOMES:
The total number of needle passes required for dural puncture. | 2012-2013
  Needle passes are defined as any forward advancement of the needle, including the first insertion and any subsequent insertion and redirection attempts. This will be assessed by two blinded observers from an anonymized video recording of the operator's hands as they perform the spinal anesthetic.
Block performance time | 2012-2013
  Block performance time, defined as the sum of the following:
  a. Time taken to establish landmarks. In the US-guided technique, this is defined as the time between first placement of the ultrasound probe on the patient and completion of the last skin marking. In the surface landmark-guided technique, this is defined as the time between first placement of the operator's hands on the patient and completion of the last skin marking.
Time taken to perform spinal anesthetic | 2012-2013
  Time taken to perform spinal anesthetic. This is defined as the period between insertion of the needle used for skin infiltration, and withdrawal of the spinal needle following injection of the

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hopspital, Toronto, Ontario, Canada